CLINICAL TRIAL: NCT02886468
Title: Determinants of Muscle - Skin Distance at the Injection Site in Patients With an Indication for the Use of Epinephrine Auto- Injector Pens
Brief Title: DEpth of EPinephrine Delivery With Auto-injectors Devices
Acronym: DEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-03-CHRMT
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Anaphylactic Shock
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ultrasound images (Experimental): ultrasound images of the anterolateral aspect of the mid-right thigh
  Interventions: Other: skin ultrasound

INTERVENTIONS:
Other: skin ultrasound

SUMMARY:
Anaphylaxis is a serious allergic reaction that is rapid in onset and may cause death. Although there are several causes of fatal anaphylaxis, food allergy is one of the most common. Epinephrine is recommended as the initial treatment of choice for anaphylaxis. A delay in epinephrine administration may contribute to an increased risk of death. Therefore, the World Allergy Organization recommends that, for the treatment of anaphylaxis, epinephrine solution be administered intramuscularly in the mid-anterolateral thigh.

In France 3 auto-injector pens are available: Anapen®, Epipen® and Jext®. For weight> 30 kg, the devices have a needle size respectively of 7.49 mm, 15.02 mm and 15.36 mm. For the weights between 15 and 30 kg needle size is 7.49 mm to 12.7 mm and Anapen® for Epipen® and Jext®.

Several studies suggest that the needle length needle is sometim

ELIGIBILITY:
Inclusion Criteria:

* a weight of over 30 kg at Baseline
* with food or an Hymenoptera venom allergy (diagnosed by skin tests or serum-specific IgE testing, requiring prescription epinephrine auto-injector pen according to European recommendations,

Exclusion Criteria:

* having a skin lesion on the lateral aspect of the thigh,
* with a known or suspected allergy to the contact gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Skin-to-muscle and muscle-to-bone distance assessment, with compression, for intramuscular injection depending on needle length of the auto-injector pen. | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Chr Metz Thionville, Metz, France

REFERENCES:
- [Derived] Lefevre S, Goetz C, Hennequin L, Zevering Y, Dinot V. Frequencies and predictors of subcutaneous and intraosseous injection with 4 epinephrine autoinjector devices. Ann Allergy Asthma Immunol. 2024 Aug;133(2):194-202.e5. doi: 10.1016/j.anai.2024.05.002. Epub 2024 May 11. PMID 38740133